CLINICAL TRIAL: NCT03356535
Title: Metabolic Signature of Healthy Lifestyle and Its Relationship With Risk of Hepatocellular Carcinoma in a Large European Cohort
Brief Title: Metabolic Signature of Healthy Lifestyle and HCC
Status: Completed | Type: Observational
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Imperial College London (Other); Danish Cancer Society (Other); University of Aarhus (Other); Centre for Research in Epidemiology and Population Health (CESP) (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); German Cancer Research Center (Other); German Institute of Human Nutrition (Other); Hellenic Health Foundation (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); ISPO Cancer Prevention and Research Institute (Unknown); Federico II University (Other); HuGeF Foundation (Unknown); Azienda Sanitaria Provinciale Ragusa (Other); University of Tromso (Other); Institut Català d'Oncologia (Other); Ministry of Health - Government of the Principality of Asturias (Other Government); Andalusian School of Public Health (Other Government); Universidad de Murcia (Other); Instituto de Salud Pública Gobierno de Navarra (Unknown); Subdirección de Salud Pública de Gipuzkoa (Unknown); Skane University Hospital (Other); Umeå University (Other); MORGEN-EPIC, Bilthoven (Unknown); Prospect-EPIC, Utrecht (Unknown); University of Oxford (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: PP201711-27
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: targeted metabolomics; multivariate statistics; metabolic signatures; partial least squares; healthy lifestyle index; EPIC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common form of liver cancer and its incidence is increasing including in regions where hepatitis infection rates are low. This trend may be the result of increases in 'unhealthy lifestyle' factors. The main aim of this study is to identify metabolic signatures associated with healthy lifestyle behaviours and to relate these signatures to risk of developing HCC to investigate whether the metabolites were of predictive utility for HCC beyond data procured from questionnaires. To address this question, we exploited data from a large European cohort (EPIC) which includes detailed questionnaire-based data as well as metabolomic data.

DETAILED DESCRIPTION:
Studies using metabolomic data have identified metabolites from several compound classes that are associated with disease-related lifestyle factors. This study identified metabolic signatures reflecting lifestyle patterns and related them to hepatocellular carcinoma (HCC) risk in the EPIC cohort. Partial Least Squares (PLS) analysis related seven modified Healthy Lifestyle Index variables (diet, BMI, physical activity, lifetime alcohol, smoking, diabetes, hepatitis) to 132 targeted serum-measured metabolites, and a liver function score in a nested study of HCC with 147 case-control pairs. The association between the resulting PLS scores and HCC risk was examined in multivariable conditional logistic regression models where odds ratios (OR) and their 95% confidence intervals (95%CI) were computed. The PLS-derived lifestyle component reflected a high propensity towards healthy behaviours. Its metabolic counterpart was positively related to the following metabolites: SM(OH) C14:1, C16:1 and C22:2, and negatively to glutamate, hexoses, and PC aaC32:1. The lifestyle and metabolomics components were inversely associated with HCC risk with OR for a 1-SD increase in scores equal to 0.49(95%CI=0.35 to 0.68) and 0.28(0.18 to 0.43).

Measuring a specific metabolites panel may identify strata of the population at higher risk for HCC and can add substantial discrimination compared to questionnaire data

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-70
* Healthy volunteers residing within defined geographical areas (where study centers are located). Different settings by centre; mostly general population with some exceptions: women of a health insurance company for teachers and school workers (France), women attending breast cancer screening (Utrecht-The Netherlands, and Florence-Italy), mainly blood donors (most centers in Italy and Spain) and a cohort consisting predominantly of vegetarians (the 'health-conscious' group in Oxford, UK)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Over 520,000 healthy men and women aged 25-85 were enrolled between 1992 and 2000 across 23 EPIC administrative centres in 10 European countries including Denmark, France, Germany, Greece, Italy, the Netherlands, Norway, Spain, Sweden, and the United Kingdom.
  This analysis focused on a nested case-control study of 147 cases of HCC and 147 matched controls with available biological samples.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Hepatocellular Carcinoma | Follow-up started at date of entry to the study and finished at date of diagnosis, death or last completed follow-up (from December 2004 up to June 2010). Cancer incidence was determined through population cancer registries or through active follow-up.
  Incident HCC cases were defined as first primary invasive tumours and identified through the 10th Revision of International Statistical Classification of Diseases, Injury and Causes of Death (ICD10) as C22.0 with morphology codes ICD-O-2 "8170/3"and "8180/3"

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Assi N, Gunter MJ, Thomas DC, Leitzmann M, Stepien M, Chajes V, Philip T, Vineis P, Bamia C, Boutron-Ruault MC, Sandanger TM, Molinuevo A, Boshuizen H, Sundkvist A, Kuhn T, Travis R, Overvad K, Riboli E, Scalbert A, Jenab M, Viallon V, Ferrari P. Metabolic signature of healthy lifestyle and its relation with risk of hepatocellular carcinoma in a large European cohort. Am J Clin Nutr. 2018 Jul 1;108(1):117-126. doi: 10.1093/ajcn/nqy074. PMID 29924298